CLINICAL TRIAL: NCT00264147
Title: A Randomized, Placebo-Controlled, Double-Blind, Multicenter, Parallel-Group, 12-Week Study to Assess the Clinically Effective Dose Range of Etoricoxib and to Assess Its Safety and Tolerability in Patients With Rheumatoid Arthritis
Brief Title: Rheumatoid Arthritis Dose Ranging Study (0663-086)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-086; 2005_077
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Results first posted 2009-07-07 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Arcoxia
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- Period I: 1 (Experimental): etoricoxib
  Interventions: Drug: etoricoxib
- Period I: 2 (Experimental): etoricoxib
  Interventions: Drug: etoricoxib
- Period I: 3 (Experimental): etoricoxib
  Interventions: Drug: etoricoxib
- Period I: 4 (Experimental): etoricoxib
  Interventions: Drug: etoricoxib
- Period I: 5 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: placebo
- Period II: 1 (Experimental): etoricoxib
  Interventions: Drug: etoricoxib
- Period II: 2 (Active Comparator): diclofenac
  Interventions: Drug: Comparator: diclofenac

INTERVENTIONS:
Drug: etoricoxib — Period I: Arm 1: etoricoxib 10 mg tablet once daily. 12 weeks of treatment.
  Arms: Period I: 1
Drug: etoricoxib — Period I: Arm 2: etoricoxib 30 mg tablet once daily. 12 weeks of treatment.
  Arms: Period I: 2
Drug: etoricoxib — Period I: Arm 3: etoricoxib 60 mg tablet once daily. 12 weeks of treatment.
  Arms: Period I: 3
Drug: etoricoxib — Period I: Arm 4: etoricoxib 90 mg tablet once daily. 12 weeks of treatment.
  Arms: Period I: 4
Drug: Comparator: placebo — Period I: Arm 5: Pbo tablet once daily. 12 weeks of treatment.
  Arms: Period I: 5
Drug: etoricoxib — Period II: Arm 1: etoricoxib 90 mg tablet once daily. 12 weeks of treatment.
  Arms: Period II: 1
Drug: Comparator: diclofenac — Period II: Arm 2: diclofenac 75 mg tablet twice daily. 12 weeks of treatment.
  Arms: Period II: 2

SUMMARY:
To assess the clinically active dose range of study medication in the treatment of patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosed rheumatoid arthritis (RA) for at least 6 months prior who is otherwise judged to be in general good health and who is currently taking nonsteroidal anti-inflammatory drugs (NSAIDS) to treat his/her RA symptoms
* Patient will need to stop taking these medications in order to participate, but can continue taking his/her other anti-rheumatic medications as long as they have been stable for certain periods of time

Exclusion Criteria:

* Patients with a disease or medical condition(s) that could worsen or interfere with the evaluation of the effectiveness of study medication are not allowed to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 761 (Actual)
Dates: Start 2006-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Greenwald M, Peloso PM, Mandel D, Soto O, Mehta A, Frontera N, Boice JA, Zhan XJ, Curtis SP. Further assessment of the clinically effective dose range of etoricoxib: a randomized, double-blinded, placebo-controlled trial in rheumatoid arthritis. Curr Med Res Opin. 2011 Oct;27(10):2033-42. doi: 10.1185/03007995.2011.614935. Epub 2011 Sep 12. PMID 21905970
- [Derived] Kvien TK, Greenwald M, Peloso PM, Wang H, Mehta A, Gammaitoni A. Do COX-2 inhibitors provide additional pain relief and anti-inflammatory effects in patients with rheumatoid arthritis who are on biological disease-modifying anti-rheumatic drugs and/or corticosteroids? Post-hoc analyses from a randomized clinical trial with etoricoxib. BMC Musculoskelet Disord. 2015 Feb 13;16:26. doi: 10.1186/s12891-015-0468-7. PMID 25886874

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 90 multicenter rheumatologists: US (71), Canada (14), Colombia (3), Switzerland (2), recruited 761 study patients from their patient pool and through advertising. First Patient In 04-Jan-2006, Last Patient Last Visit 26-Mar-2008.
Pre-assignment Details: Patients must have taken Non Steroidal Anti-inflammatory Drugs (NSAIDs) at a therapeutic labeled dose on a regular basis and demonstrated a clinical response in the past and at screening. Following a protocol-specified "washout," patients must have demonstrated disease activity and worsening in symptoms of Rheumatoid Arthritis from the screening.
Groups:
- Placebo: Treatment I: Placebo orally once daily
- Etoricoxib 10 mg: Treatment I: Etoricoxib 10 mg orally once daily
- Etoricoxib 30 mg: Treatment I: Etoricoxib 30 mg orally once daily
- Etoricoxib 60 mg: Treatment I: Etoricoxib 60 mg orally once daily
- Etoricoxib 90 mg: Treatment I and II: Etoricoxib 90 mg orally once daily
- Diclofenac 150 mg (Treatment II): Treatment II: Diclofenac 75 mg orally twice daily
Period: Treatment I Period
Arm/Group | Placebo | Etoricoxib 10 mg | Etoricoxib 30 mg | Etoricoxib 60 mg | Etoricoxib 90 mg | Diclofenac 150 mg (Treatment II)
Started | 161 | 154 | 151 | 140 | 155 | 0
Completed | 63 (Randomized to Treatment I period and remained on Treatment I period during course of study) | 71 (Randomized to Treatment I period and remained on Treatment I period during course of study) | 74 (Randomized to Treatment I period and remained on Treatment I period during course of study) | 68 (Randomized to Treatment I period and remained on Treatment I period during course of study) | 99 (Randomized to Treatment I period and remained on Treatment I period during course of study) | 0
Not Completed | 98 | 83 | 77 | 72 | 56 | 0
Not completed — Adverse Event | 3 | 6 | 3 | 5 | 7 | 0
Not completed — Laboratory Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 6 | 2 | 8 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 2 | 2 | 0
Not completed — Patient out of town for an extended time | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Unblinded due to Serious Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Reassigned to Treatment II Period | 84 | 72 | 65 | 63 | 45 | 0
Period: Treatment II Period
Arm/Group | Placebo | Etoricoxib 10 mg | Etoricoxib 30 mg | Etoricoxib 60 mg | Etoricoxib 90 mg | Diclofenac 150 mg (Treatment II)
Started | 0 | 0 | 0 | 0 | 180 (Etoricoxib 10 mg (38), 30 mg (28), 60 mg (33), 90 mg (45) and placebo (36) reassigned to 90 mg (180)) | 149 (Etoricoxib 10 mg (34), 30 mg (37), 60 mg (29), and placebo (49) reassigned to diclofenac (149))
Completed | 0 | 0 | 0 | 0 | 147 | 116
Not Completed | 0 | 0 | 0 | 0 | 33 | 33
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 9 | 9
Not completed — Laboratory Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 20 | 19
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 2
Not completed — Pre-scheduled total hip replacement | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Etoricoxib 90 mg: Treatment I: Etoricoxib 90 mg orally once daily
- Total: Total of all reporting groups
Arm/Group | Placebo | Etoricoxib 10 mg | Etoricoxib 30 mg | Etoricoxib 60 mg | Etoricoxib 90 mg | Total
Number analyzed (Participants) | 161 | 154 | 151 | 140 | 155 | 761
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (11.80) | 58.7 (11.92) | 56.2 (11.17) | 57.7 (10.96) | 54.9 (12.54) | 57.0 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 117 | 126 | 112 | 122 | 613
  Male | 25 | 37 | 25 | 28 | 33 | 148
American Rheumatism Association Functional Class [Number; unit: Participants] — Class I: Completely able to perform usual activities of daily living (self care, vocational, and avocational), Class II: Able to perform usual self-care and vocational activities, but limited in avocational activities, Class III: Able to perform usual self-care activities, but limited in vocational and avocational activities
  Participants
    Class I | 44 | 49 | 49 | 41 | 38 | 221
    Class II | 102 | 83 | 83 | 73 | 98 | 439
    Class III | 15 | 22 | 19 | 26 | 19 | 101
Corticosteroid User [Number; unit: Participants]
  Yes | 50 | 50 | 42 | 41 | 49 | 232
  No | 111 | 104 | 109 | 99 | 106 | 529
Disease Modifying Antirheumatic Drug User [Number; unit: Participants]
  Yes | 133 | 129 | 122 | 114 | 131 | 629
  No | 28 | 25 | 29 | 26 | 24 | 132
Disease Modifying Antirheumatic Drug or Corticosteroid User [Number; unit: Participants]
  Yes | 139 | 134 | 126 | 119 | 136 | 654
  No | 22 | 20 | 25 | 21 | 19 | 107
Methotrexate User [Number; unit: Participants]
  Yes | 99 | 91 | 96 | 93 | 93 | 472
  No | 62 | 63 | 55 | 47 | 62 | 289
Race/Ethnicity [Number; unit: participants]
  Asian | 1 | 0 | 1 | 1 | 1 | 4
  Black | 5 | 8 | 3 | 7 | 6 | 29
  White | 114 | 106 | 121 | 96 | 112 | 549
  Hispanic | 41 | 39 | 25 | 34 | 36 | 175
  Native American | 0 | 0 | 1 | 2 | 0 | 3
  Indian | 0 | 1 | 0 | 0 | 0 | 1
Rheumatoid Factor [Number; unit: Participants]
  Positive | 120 | 117 | 121 | 120 | 121 | 599
  Negative | 40 | 37 | 30 | 20 | 34 | 161
  Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Smoking Status [Number; unit: Participants]
  Current | 27 | 28 | 29 | 23 | 22 | 129
  Ex-User | 53 | 46 | 42 | 39 | 40 | 220
  Non-User | 81 | 80 | 80 | 78 | 93 | 412
Body Weight [Mean (Standard Deviation); unit: Kilograms] | 76.42 (16.54) | 76.12 (18.48) | 77.36 (20.00) | 75.72 (19.54) | 77.97 (18.61) | 76.73 (18.58)
Duration of Rheumatoid Arthritis (Years) [Mean (Standard Deviation); unit: Years] | 10.0 (9.78) | 10.1 (9.76) | 11.2 (8.40) | 10.3 (10.18) | 9.9 (9.98) | 10.3 (9.62)
Height [Mean (Standard Deviation); unit: Centimeters] | 161.93 (9.71) | 163.63 (8.55) | 164.57 (9.13) | 162.96 (9.22) | 163.49 (10.04) | 163.30 (9.37)
Investigator Global Assessment of Disease Activity (0 to 4 - Likert Scale) [Mean (Standard Deviation); unit: units on a scale] — (0 to 4 - Likert Scale) 0=Very Well, 1=Well, 2=Fair, 3=Poor, 4=Very Poor
  units on a scale | 2.71 (0.61) | 2.71 (0.67) | 2.75 (0.66) | 2.69 (0.63) | 2.73 (0.65) | 2.72 (0.64)
Patient Global Assessment of Disease Activity (0-To- 100 Millimeter Visual Analog Scale) [Mean (Standard Deviation); unit: units on a scale] — (0- to 100-mm Visual Analog Scale) 0 mm= No pain, 100 mm= Extreme pain
  units on a scale | 66.08 (18.67) | 69.28 (19.37) | 66.56 (20.47) | 66.60 (19.58) | 65.42 (18.45) | 66.79 (19.30)
Patient Global Assessment of Pain (0- To- 100-mm Visual Analog Scale) [Mean (Standard Deviation); unit: units on a scale] — (0- to 100-mm Visual Analog Scale) 0 mm= No pain, 100 mm= Extreme pain
  units on a scale | 72.66 (16.03) | 72.42 (17.32) | 70.95 (16.67) | 69.54 (18.24) | 71.08 (17.55) | 71.38 (17.14)
Swollen Joint Count (Out of 66 Joints) [Mean (Standard Deviation); unit: Number of Swollen Joints] | 16.05 (9.79) | 17.75 (10.86) | 16.74 (10.11) | 15.79 (9.40) | 16.30 (10.05) | 16.53 (10.06)
Tender Joint Count (Out of 68 Joints) [Mean (Standard Deviation); unit: Number of Tender Joints] | 26.91 (14.17) | 28.33 (15.42) | 27.19 (14.97) | 26.76 (14.37) | 27.25 (16.11) | 27.30 (15.00)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Met the ACR20 Responder Index Criteria
Description: Proportion of Patients Who Met the American College of Rheumatology Response Index (20%) Criteria (ACR20) (Based on the Time-Weighted Average Responses of the 12-Week Treatment I Period and Completed the Treatment I Period) (All Patients-Treated Population)
Time Frame: 12 weeks
Population: All-Patients-Treated Population
Measure: Number; unit: Proportion of Patients
Arm/Group | Placebo | Etoricoxib 10 mg | Etoricoxib 30 mg | Etoricoxib 60 mg | Etoricoxib 90 mg
Number analyzed (Participants) | 161 | 154 | 151 | 140 | 155
Proportion of Patients | 28.57 | 35.06 | 37.75 | 38.57 | 47.10
Statistical Analysis 1: Comparison: Placebo vs Etoricoxib 10 mg vs Etoricoxib 30 mg vs Etoricoxib 60 mg vs Etoricoxib 90 mg; Test type: Superiority or Other; p < 0.001, Cochran-Armitage trend test — Overall alpha=0.05 for multiple comparisons with a step-down procedure (p-values subsequent to the first non-significant p-value were not reported); A step-down procedure and Abelson-Tukey scaling were used for the trend test
Statistical Analysis 2: Comparison: Placebo vs Etoricoxib 10 mg vs Etoricoxib 30 mg vs Etoricoxib 60 mg; Test type: Superiority or Other; p = 0.057, Cochran-Armitage trend test — [p-value comment as in outcome 1, analysis 1]; A step-down procedure and Abelson-Tukey scaling were used for the trend test
Statistical Analysis 3: Comparison: Placebo vs Etoricoxib 90 mg; Test type: Superiority or Other; difference in percentage of patients = 18.53, 95% CI [7.84 to 28.65] — CI based on the Wilson's score method
Statistical Analysis 4: Comparison: Placebo vs Etoricoxib 60 mg; Test type: Superiority or Other; difference in percentage of patients = 10.00, 95% CI [-0.66 to 20.46] — CI based on the Wilson's score method
Statistical Analysis 5: Comparison: Placebo vs Etoricoxib 30 mg; Test type: Superiority or Other; difference in percentage of patients = 9.18, 95% CI [-1.25 to 19.39] — CI based on the Wilson's score method
Statistical Analysis 6: Comparison: Placebo vs Etoricoxib 10 mg; Test type: Superiority or Other; difference in percentage of patients = 6.49, 95% CI [-3.76 to 16.61] — CI based on the Wilson's score method

2. Secondary Outcome: Tender Joint Count (Out of 68 Joints) Time-Weighted Average Change From Baseline (Flare/Randomization Visit) in the 12-Week Treatment Period (All Patients-Treated Population)
Time Frame: Time-weighted average change from baseline across Weeks 2, 7, and 12
Population: All-Patients-Treatment Population
Measure: Mean (Standard Deviation); unit: Tender Joint Count
Arm/Group | Placebo | Etoricoxib 10 mg | Etoricoxib 30 mg | Etoricoxib 60 mg | Etoricoxib 90 mg
Number analyzed (Participants) | 157 | 148 | 146 | 138 | 148
Tender Joint Count | -8.13 (9.55) | -11.01 (13.07) | -10.96 (11.00) | -9.56 (11.85) | -12.06 (11.22)
Statistical Analysis 1: Comparison: Placebo vs Etoricoxib 10 mg vs Etoricoxib 30 mg vs Etoricoxib 60 mg vs Etoricoxib 90 mg; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on a trend test with a step-down procedure and Abelson-Tukey scaling
Statistical Analysis 2: Comparison: Placebo vs Etoricoxib 10 mg vs Etoricoxib 30 mg vs Etoricoxib 60 mg; Test type: Superiority or Other; p = 0.221, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on a trend test with a step-down procedure and Abelson-Tukey scaling
Statistical Analysis 3: Comparison: Placebo vs Etoricoxib 90 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -4.06, 95% CI [-6.44 to -1.68]
Statistical Analysis 4: Comparison: Placebo vs Etoricoxib 60 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -1.49, 95% CI [-3.91 to 0.93]
Statistical Analysis 5: Comparison: Placebo vs Etoricoxib 30 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -2.74, 95% CI [-5.13 to -0.35]
Statistical Analysis 6: Comparison: Placebo vs Etoricoxib 10 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -2.50, 95% CI [-4.88 to -0.12]

3. Secondary Outcome: Swollen Joint Count (Out of 66 Joints) Time-Weighted Average Change From Baseline (Flare/Randomization Visit) in the 12-Week Treatment Period (All Patients-Treated Population)
Time Frame: Time-weighted average change from baseline across Weeks 2, 7, and 12
Population: All-Patients-Treatment Population
Measure: Mean (Standard Deviation); unit: Swollen Joint Count
Arm/Group | Placebo | Etoricoxib 10 mg | Etoricoxib 30 mg | Etoricoxib 60 mg | Etoricoxib 90 mg
Number analyzed (Participants) | 157 | 148 | 146 | 138 | 148
Swollen Joint Count | -5.39 (7.34) | -6.58 (8.11) | -6.91 (7.27) | -6.25 (7.48) | -7.77 (7.17)
Statistical Analysis 1: Comparison: Placebo vs Etoricoxib 10 mg vs Etoricoxib 30 mg vs Etoricoxib 60 mg vs Etoricoxib 90 mg; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on a trend test with a step-down procedure and Abelson-Tukey scaling
Statistical Analysis 2: Comparison: Placebo vs Etoricoxib 10 mg vs Etoricoxib 30 mg vs Etoricoxib 60 mg; Test type: Superiority or Other; p = 0.125, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on a trend test with a step-down procedure and Abelson-Tukey scaling
Statistical Analysis 3: Comparison: Placebo vs Etoricoxib 90 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -2.24, 95% CI [-3.64 to -0.84]
Statistical Analysis 4: Comparison: Placebo vs Etoricoxib 60 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -1.02, 95% CI [-2.44 to 0.41]
Statistical Analysis 5: Comparison: Placebo vs Etoricoxib 30 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -1.22, 95% CI [-2.63 to 0.18]
Statistical Analysis 6: Comparison: Placebo vs Etoricoxib 10 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.49, 95% CI [-1.89 to 0.91]

4. Secondary Outcome: Patient Global Assessment of Disease Activity (0- to 100-mm Visual Analog Scale) Time Weighted Average Change From Baseline (Flare/Randomization Visit) in the 12-Week Treatment I Period (All Patients-Treated Population)
Description: 0-mm indicates very well, 100-mm indicates very poor.
Time Frame: Time-weighted average change from baseline across Weeks 2, 7, and 12
Population: All Patients-Treated Population
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Etoricoxib 10 mg | Etoricoxib 30 mg | Etoricoxib 60 mg | Etoricoxib 90 mg
Number analyzed (Participants) | 155 | 144 | 141 | 134 | 144
Units on a Scale | -12.32 (25.66) | -19.90 (23.61) | -21.12 (24.47) | -21.49 (26.71) | -25.75 (25.71)
Statistical Analysis 1: Comparison: Placebo vs Etoricoxib 10 mg vs Etoricoxib 30 mg vs Etoricoxib 60 mg vs Etoricoxib 90 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on a trend test with a step-down procedure and Abelson-Tukey scaling
Statistical Analysis 2: Comparison: Placebo vs Etoricoxib 10 mg vs Etoricoxib 30 mg vs Etoricoxib 60 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on a trend test with a step-down procedure and Abelson-Tukey scaling
Statistical Analysis 3: Comparison: Placebo vs Etoricoxib 10 mg vs Etoricoxib 30 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on a trend test with a step-down procedure and Abelson-Tukey scaling
Statistical Analysis 4: Comparison: Placebo vs Etoricoxib 10 mg; Test type: Superiority or Other; p = 0.023, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on a trend test with a step-down procedure and Abelson-Tukey scaling
Statistical Analysis 5: Comparison: Placebo vs Etoricoxib 90 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -14.16, 95% CI [-19.38 to -8.95]
Statistical Analysis 6: Comparison: Placebo vs Etoricoxib 60 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -9.21, 95% CI [-14.52 to -3.90]
Statistical Analysis 7: Comparison: Placebo vs Etoricoxib 30 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -8.87, 95% CI [-14.11 to -3.63]
Statistical Analysis 8: Comparison: Placebo vs Etoricoxib 10 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -6.05, 95% CI [-11.27 to -0.83]

5. Secondary Outcome: Investigator Global Assessment of Disease Activity (0- to 4-Likert Scale) Time Weighted Average Change From Baseline (Flare/Randomization Visit) in the 12-Week Treatment I Period (All Patients-Treated Population)
Description: 0 indicates very well, 4 indicates very poor.
Time Frame: Time-weighted average change from baseline across Weeks 2, 7, and 12
Population: All-Patients-Treatment Population
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Etoricoxib 10 mg | Etoricoxib 30 mg | Etoricoxib 60 mg | Etoricoxib 90 mg
Number analyzed (Participants) | 157 | 148 | 146 | 138 | 148
Units on a Scale | -0.68 (1.06) | -0.93 (0.94) | -1.09 (1.01) | -1.01 (0.94) | -1.24 (0.94)
Statistical Analysis 1: Comparison: Placebo vs Etoricoxib 10 mg vs Etoricoxib 30 mg vs Etoricoxib 60 mg vs Etoricoxib 90 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on a trend test with a step-down procedure and Abelson-Tukey scaling
Statistical Analysis 2: Comparison: Placebo vs Etoricoxib 10 mg vs Etoricoxib 30 mg vs Etoricoxib 60 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on a trend test with a step-down procedure and Abelson-Tukey scaling
Statistical Analysis 3: Comparison: Placebo vs Etoricoxib 10 mg vs Etoricoxib 30 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on a trend test with a step-down procedure and Abelson-Tukey scaling
Statistical Analysis 4: Comparison: Placebo vs Etoricoxib 10 mg; Test type: Superiority or Other; p = 0.018, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on a trend test with a step-down procedure and Abelson-Tukey scaling
Statistical Analysis 5: Comparison: Placebo vs Etoricoxib 90 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.56, 95% CI [-0.77 to -0.35]
Statistical Analysis 6: Comparison: Placebo vs Etoricoxib 60 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.34, 95% CI [-0.55 to -0.13]
Statistical Analysis 7: Comparison: Placebo vs Etoricoxib 30 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.40, 95% CI [-0.61 to -0.19]
Statistical Analysis 8: Comparison: Placebo vs Etoricoxib 10 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.25, 95% CI [-0.46 to -0.04]

6. Secondary Outcome: Patient Global Assessment of Pain (0- to 100-mm Visual Analog Scale) Time Weighted Average Change From Baseline (Flare/Randomization Visit) in the 12-Week Treatment I Period (All Patients-Treated Population)
Description: 0-mm indicates very well, 100-mm indicates very poor.
Time Frame: Time-weighted average change from baseline across Weeks 2, 7, and 12
Population: All-Patients-Treated Population
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Etoricoxib 10 mg | Etoricoxib 30 mg | Etoricoxib 60 mg | Etoricoxib 90 mg
Number analyzed (Participants) | 157 | 148 | 146 | 137 | 148
Units on a Scale | -17.44 (23.42) | -21.95 (22.87) | -22.75 (23.86) | -22.25 (26.58) | -31.07 (24.18)
Statistical Analysis 1: Comparison: Placebo vs Etoricoxib 10 mg vs Etoricoxib 30 mg vs Etoricoxib 60 mg vs Etoricoxib 90 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on a trend test with a step-down procedure and Abelson-Tukey scaling
Statistical Analysis 2: Comparison: Placebo vs Etoricoxib 10 mg vs Etoricoxib 30 mg vs Etoricoxib 60 mg; Test type: Superiority or Other; p = 0.018, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on a trend test with a step-down procedure and Abelson-Tukey scaling
Statistical Analysis 3: Comparison: Placebo vs Etoricoxib 10 mg vs Etoricoxib 30 mg; Test type: Superiority or Other; p = 0.017, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on a trend test with a step-down procedure and Abelson-Tukey scaling
Statistical Analysis 4: Comparison: Placebo vs Etoricoxib 10 mg; Test type: Superiority or Other; p = 0.080, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Based on a trend test with a step-down procedure and Abelson-Tukey scaling
Statistical Analysis 5: Comparison: Placebo vs Etoricoxib 90 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -14.44, 95% CI [-19.62 to -9.26]
Statistical Analysis 6: Comparison: Placebo vs Etoricoxib 60 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -6.22, 95% CI [-11.52 to -0.92]
Statistical Analysis 7: Comparison: Placebo vs Etoricoxib 30 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -6.32, 95% CI [-11.53 to -1.12]
Statistical Analysis 8: Comparison: Placebo vs Etoricoxib 10 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -4.63, 95% CI [-9.81 to 0.55]

ADVERSE EVENTS:
Groups:
- Placebo Treatment I Period: Treatment I: Placebo orally once daily
- Etoricoxib 10 mg Treatment I Period: Treatment I: Etoricoxib 10 mg orally once daily
- Etoricoxib 30 mg Treatment I Period: Treatment I: Etoricoxib 30 mg orally once daily
- Etoricoxib 60 mg Treatment I Period: Treatment I: Etoricoxib 60 mg orally once daily
- Etoricoxib 90 mg Treatment I Period: Treatment I: Etoricoxib 90 mg orally once daily
- Etoricoxib 90 mg Treatment II Period: Treatment II: Etoricoxib 90 mg orally once daily
- Diclofenac 150 mg Treatment II Period: Treatment II: Diclofenac 75 mg orally twice daily
Arm/Group | Placebo Treatment I Period | Etoricoxib 10 mg Treatment I Period | Etoricoxib 30 mg Treatment I Period | Etoricoxib 60 mg Treatment I Period | Etoricoxib 90 mg Treatment I Period | Etoricoxib 90 mg Treatment II Period | Diclofenac 150 mg Treatment II Period
Serious Adverse Events (participants affected / at risk) | 0 | 1 | 4 | 1 | 5 | 3 | 3
Other Adverse Events (participants affected / at risk) | 28 | 19 | 29 | 37 | 39 | 25 | 30
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Placebo Treatment I Period | Etoricoxib 10 mg Treatment I Period | Etoricoxib 30 mg Treatment I Period | Etoricoxib 60 mg Treatment I Period | Etoricoxib 90 mg Treatment I Period | Etoricoxib 90 mg Treatment II Period | Diclofenac 150 mg Treatment II Period
Coronary Artery Disease (Cardiac disorders) | 0/161 | 0/154 | 1/151 | 0/140 | 0/155 | 0/180 | 0/149
Myocardial Infarction (Cardiac disorders) | 0/161 | 0/154 | 1/151 | 0/140 | 0/155 | 0/180 | 0/149
Gastritis (Gastrointestinal disorders) | 0/161 | 0/154 | 1/151 | 0/140 | 0/155 | 0/180 | 0/149
Ileus Paralytic (Gastrointestinal disorders) | 0/161 | 0/154 | 1/151 | 0/140 | 0/155 | 0/180 | 0/149
Small Intestinal Obstruction (Gastrointestinal disorders) | 0/161 | 0/154 | 0/151 | 0/140 | 1/155 | 0/180 | 0/149
Cellulitis (Infections and infestations) | 0/161 | 0/154 | 0/151 | 0/140 | 1/155 | 0/180 | 0/149
Erysipelas (Infections and infestations) | 0/161 | 0/154 | 1/151 | 0/140 | 0/155 | 0/180 | 0/149
Accidental Overdose (Injury, poisoning and procedural complications) | 0/161 | 0/154 | 0/151 | 0/140 | 0/155 | 0/180 | 1/149
Dislocation Of Joint Prosthesis (Injury, poisoning and procedural complications) | 0/161 | 0/154 | 0/151 | 0/140 | 1/155 | 0/180 | 0/149
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0/161 | 0/154 | 0/151 | 0/140 | 0/155 | 1/180 | 0/149
Heat Exhaustion (Injury, poisoning and procedural complications) | 0/161 | 0/154 | 0/151 | 0/140 | 1/155 | 0/180 | 0/149
Blood Creatinine Increased (Investigations) | 0/161 | 0/154 | 0/151 | 1/140 | 0/155 | 0/180 | 0/149
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0/161 | 0/154 | 1/151 | 0/140 | 0/155 | 0/180 | 0/149
Malignant Melanoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/161 | 0/154 | 0/151 | 0/140 | 0/155 | 0/180 | 1/149
Depression (Psychiatric disorders) | 0/161 | 0/154 | 0/151 | 0/140 | 1/155 | 0/180 | 0/149
Obsessive-Compulsive Disorder (Psychiatric disorders) | 0/161 | 0/154 | 0/151 | 0/140 | 0/155 | 0/180 | 1/149
Ovarian Cyst (Reproductive system and breast disorders) | 0/161 | 0/154 | 0/151 | 0/140 | 0/155 | 1/180 | 0/149
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0/161 | 0/154 | 1/151 | 0/140 | 0/155 | 0/180 | 0/149
Dermatitis (Skin and subcutaneous tissue disorders) | 0/161 | 0/154 | 0/151 | 0/140 | 0/155 | 1/180 | 0/149
Hypertension (Vascular disorders) | 0/161 | 1/154 | 0/151 | 0/140 | 0/155 | 0/180 | 0/149
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Placebo Treatment I Period | Etoricoxib 10 mg Treatment I Period | Etoricoxib 30 mg Treatment I Period | Etoricoxib 60 mg Treatment I Period | Etoricoxib 90 mg Treatment I Period | Etoricoxib 90 mg Treatment II Period | Diclofenac 150 mg Treatment II Period
Abdominal Pain (Gastrointestinal disorders) | 0/161 | 0/154 | 0/151 | 0/140 | 1/155 | 0/180 | 3/149
Abdominal Pain Upper (Gastrointestinal disorders) | 2/161 | 1/154 | 1/151 | 3/140 | 2/155 | 0/180 | 2/149
Constipation (Gastrointestinal disorders) | 0/161 | 1/154 | 5/151 | 3/140 | 2/155 | 1/180 | 1/149
Diarrhoea (Gastrointestinal disorders) | 3/161 | 4/154 | 2/151 | 8/140 | 7/155 | 4/180 | 6/149
Dyspepsia (Gastrointestinal disorders) | 5/161 | 2/154 | 1/151 | 3/140 | 6/155 | 2/180 | 4/149
Nausea (Gastrointestinal disorders) | 2/161 | 2/154 | 2/151 | 3/140 | 3/155 | 0/180 | 2/149
Oedema Peripheral (General disorders) | 1/161 | 2/154 | 2/151 | 5/140 | 1/155 | 6/180 | 4/149
Nasopharyngitis (Infections and infestations) | 1/161 | 4/154 | 0/151 | 1/140 | 4/155 | 2/180 | 1/149
Sinusitis (Infections and infestations) | 3/161 | 1/154 | 0/151 | 1/140 | 4/155 | 2/180 | 1/149
Upper Respiratory Tract Infection (Infections and infestations) | 4/161 | 0/154 | 4/151 | 1/140 | 2/155 | 4/180 | 7/149
Urinary Tract Infection (Infections and infestations) | 1/161 | 1/154 | 3/151 | 0/140 | 0/155 | 2/180 | 1/149
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 3/161 | 1/154 | 3/151 | 4/140 | 2/155 | 1/180 | 3/149
Dizziness (Nervous system disorders) | 1/161 | 1/154 | 2/151 | 4/140 | 6/155 | 0/180 | 1/149
Headache (Nervous system disorders) | 6/161 | 4/154 | 5/151 | 8/140 | 5/155 | 2/180 | 0/149
Cough (Respiratory, thoracic and mediastinal disorders) | 1/161 | 1/154 | 0/151 | 3/140 | 2/155 | 0/180 | 1/149
Hypertension (Vascular disorders) | 0/161 | 2/154 | 3/151 | 6/140 | 5/155 | 6/180 | 1/149

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.